CLINICAL TRIAL: NCT03229603
Title: A Pilot Study on HPV and Cervical Cancer Screening in Mumbai
Acronym: HPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: University of Arizona (Other)
Responsible Party: Principal Investigator, Gauravi Ashish Mishra, Professor and Physician, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TMHPO1763
Record Dates: First submitted 2017-04-18; First posted 2017-07-25 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-07

CONDITIONS: HPV Infection
Keywords: HPV infection and Cervical cancer
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cluster of 3000 women (Other): Cluster will be selected from an existing cervical, breast, and oral cancer screening program in Mumbai, India and its surrounding semi-urban and rural areas.
  Interventions: Other: Cluster of 3000 women

INTERVENTIONS:
Other: Cluster of 3000 women — An evaluation of the feasibility, reach, adoption and implementation of a cervical cancer screening program where we diagnose HPV using the GeneXpert point of care testing kit prior to VIA and cryotherapy.

SUMMARY:
The Study goals are to test feasibility and acceptability of point of care HPV testing with 227 women already accessing an existing cancer screening program in Mumbai, India. Describe HPV infection types in women screened. Compare if the quality of HPV clinician-collected and self-collected samples are equally efficient to detect HPV and cervical cancer precursor lesions. Compare the agreement between HPV GeneXpert and HPV HC2 test on the clinician-collected sample

DETAILED DESCRIPTION:
In this pilot study, Investigators will assess the feasibility and acceptability of point of care HPV testing in an existing SVA program. There is no control group since neither the efficacy nor effectiveness is to be tested. In the pilot study the screen positive women will be referred to the Tata Memorial Hospital for further diagnostic work-up to restrict the programme logistics. While in the main study, Colposcopy and Cryotherapy will be conducted at the community level. The evaluation framework will be based on a robust D&I model called REAIM.

i.TMH staff will hold health camps to mobilize women to attend. Providers already trained in the TMH outreach program will identify women eligible for screening. After obtaining the consent, the medical social worker will collect baseline data and record the results of the GeneXpert HPV testing on self sample and health care provider collected sample.

Data Collection:

ii. Quantitative data: Data will be collected in-person by the Medical Social worker. De-identified data will be uploaded to Own Cloud, a file-sharing program in the University of Arizona, College of Nursing.

ii. Qualitative data: There will be a discussion on cultural appropriateness and possible adjustments to the procedures based on the healthcare providers' experiences with a small subset of the 227 women already screened. Between one to two focus groups will be conducted by the study investigators with assistance from local staff with a subset of women, separately to qualitatively assess acceptability of HPV testing using GeneXpert.

The focus group discussions with women participants will be audio-recorded and transcribed verbatim. The moderator will be guided by a semi-structured set of questions to facilitate discussion, and will specifically probe to elicit distinctive/ unusual behaviors or symptoms related to the program, screening and HPV testing.

In keeping with standards for objective evaluation, Dr. Menon or Kue will conduct a focus group discussion with Medical Social workers at the end of the study period for program evaluation (i.e., acceptability, potential changes in delivery, etc.). Discussions will be recorded by a note-taker, not previously associated with the study.

Given the small numbers, a think-aloud group, in a question and answer format with a note-taker to record the main points will be simply conducted with the providers. Both the facilitator and note-taker will not be among TMH staff as this may introduce bias to the conversation.

iii: Training of TMH staff to use GeneXpert: Personnel from the India office of Cepheid will train providers on how to use GeneXpert using standardized training protocols. The quality of the self- collected sample will be compared to the quality of the provider collected sample (by running two separate GeneXpert tests on each sample) to establish the feasibility of self-sampling.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 30 to 55 years (the age when screening for HPV and cervical cancer is recommended) who participate in the TMH cancer screening outreach program.

Exclusion Criteria:

* Women with a known diagnosis of cancer, any other terminal diagnosis, or who are pregnant

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 227 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The feasibility of HPV testing as a single visit approach will be summarized using the appropriate descriptive statistics. | 3 months
  This will be predominantly for counts and percentages for categorical variables (e.g., number of women screened, number of women with incomplete self-collected specimens). In addition to the numbers of participants, the notes from the providers' debriefing regarding culturally appropriateness of HPV testing will be considered.

SECONDARY OUTCOMES:
Overall agreement between clinician-collected versus self-collected samples will be compared using pairwise t tests | 3 months
  For all pairwise comparisons, the agreement will be estimated with the kappa statistic and corresponding 95% confidence intervals. McNemar's test shall be used to detect significant differences in the discordant results (p<0.05), indicating systematic differences by assay or sample type in the detection of HPV.
The focus group data will be analyzed using constant comparative data analysis to identify thematic components and sub-themes. | 3 months
  The research team will conduct a content analysis taking the following approach set forth by Huberman and Miles.
The HPV GeneXpert by health care provider and HPV HC2 samples by health care provider will be compared to study the agreement rates. | 3 months
  For all pairwise comparisons, the agreement will be estimated with the kappa statistic and corresponding 95% confidence intervals. McNemar's test shall be used to detect significant differences in the discordant results (p<0.05), indicating systematic differences by assay or sample type in the detection of HPV.
Documentation of six different genotypes/ genotype families of HPV from cervical tissue samples, which will inform the development of HPV vaccinations specific to the strains of HPV in India. | 3 months
  The prevalence and distribution of HPV genotypes in Indian women with cervical cancer and the trends in HPV infections will be summarized using the appropriate descriptive statistics.
Probe for perceptions about self-collection of vaginal samples to describe acceptability of this process. | 3 months
  Mainly descriptive statistics in percentage, numbers and description
Fit a predictive model of HPV infection(s). | 3 months
  This will be predicted by sexual behavior, sociodemographic and clinical characteristics of the women screened, controlling for the two screening sites. A positive intra-class correlation (ICC) is expected among participants at the same screening site due to commonalities in selection, exposure, mutual interaction, or a combination of those factors. We will fit Linear Mixed Models (LMMs) and Generalized Linear Mixed Models (GLMMs) to account for various levels of correlation among participants (also known as a "mixed-model ANCOVA" (Brown, 2009). We will fit these models using SAS PROC MIXED and GLIMMIX, Version 9.3.

CONTACTS AND LOCATIONS:
Overall Officials: Gauravi A Mishra, M.D PSM, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided